CLINICAL TRIAL: NCT01644747
Title: tDCS as an add-on Treatment for Resistant Major Depression in Uni- or Bipolar Patients: a Randomized, Double-blind, Placebo Controlled Study
Brief Title: tDCS as an add-on Treatment for Resistant Major Depression in Uni- or Bipolar Patients
Acronym: STICODEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); University Hospital, Grenoble (Other); CH Le Vinatier - Service de Psychiatrie (Dr Emmanuel POULET) (Unknown); Rennes University Hospital (Other); EPS Ville-Evrard - Unité de Recherche Clinique (Dr Dominique JANUEL) (Unknown); Hôpital Civil de Strasbourg - Service de Psychiatrie (Pr G.Bertschy) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N/2011/60
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Resistant Depression; Moods Disorders; Unipolar Depression; Bipolar Disorder
Keywords: Resistant Depression; Moods disorders; Unipolar depression; Bipolar disorder; tDCS
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active tDCS (Active Comparator): a group named G1 and treated by medication with SSRIs (Selective Serotonin Reuptake Inhibitors) or SNRIs (Serotonine-Norepinephrine Reuptake Inhibitors) for 48 unipolar patients or with Lithium for 12 bipolar patients stabilized for at least 4 months and 10 sessions of active anodal tDCS at 2 sessions per day (1 morning and 1 afternoon with a gap of 3h) for 5 days with an electric current 2 mA.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS) (Eldith DC NeuroConn Stimulator)
- sham tDCS (Sham Comparator): a group named G2 and treated by medication with SSRIs or SNRIs for 48 unipolar patients or with Lithium for 12 bipolar patients stabilized for at least 4 months and sham tDCS.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS) (Eldith DC NeuroConn Stimulator)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) (Eldith DC NeuroConn Stimulator) — After locating the left DLPFC, ttt with active anodal tDCS with a current of 2 mA or sham over the left DLPFC will be directed by 30-minute session. Treatment will occur 2 sessions per day during 5 days per week. Subjects will be monitored during tDCS for any side effects or adverse events.
  Other Names: EldithDC-NeuroConn Stimulator (NeuroConn Gmbh, Ilmenau, Germany)

SUMMARY:
The aim is to investigate the effect of transcranial Direct Current Stimulation (tDCS) applied at the anodal left CDLPF of patients with resistant depression compared to patients treated with conventional therapy. The tDCS is used in add-on drug treatment in resistant depression stabilized for 4 weeks (antidepressant as SSRIs (Selective Serotonin Reuptake Inhibitors) or SNRIs (Serotonine-Norepinephrine Reuptake Inhibitors) for unipolar patients and lithium for bipolar patients). The delay of 4 weeks is a minimum to observe a non-response. Moreover, in term of ethical point of view, it's difficult to wait 6 to 8 weeks to observe the non-response to treatment.

This is a randomized 2-arm parallel, double blind study comparing 2 groups of 60 patients (48 unipolar plus 12 bipolar patients per group. Patients will be selected in the psychiatric department of the University Hospital of different centers and the two groups are matched for age (+/- 5 years), gender and depression diagnosis (unipolar vs bipolar).

After giving informed consent, patients will be evaluated by a psychiatrist using the Hamilton Depression Rating Scale (HDRS), Montgomery Asberg Depression Rating Scale (MADRS), the STAI and Beck Depression Inventory (BDI) and for bipolar patient only, by the Young Mania Rating Scale (YMRS). The complete assessment takes 50 minutes. A neuropsychologist assessment will be also realized during 20 minutes using the Crossing of Test (COT), the Trail Making Test (TMT), the Isaacs Set Test (IST) and the Cardebat fluency Task.

After locating the left DLPFC, treatment with active tDCS with a current of 2 mA or sham will be directed by 30-minute session. A psychometric assessment will be conducted again at the end of treatment week and 4, 12 and finally 24 weeks after stopping treatment. The neuropsychologist assessment will be conducted again 4 weeks after the end of treatment. Scales of comfort and acceptability will also be proposed to the patient to determine whether any gene is caused by this treatment.

These people will be recruited on a voluntary basis, after notification and consent in the 6 research centers. This study was conducted over a period of 36 months.

This study was supporting by a grant from the French Hospital Program of Clinical Reseach (PHRC N/2011-60-2011-A01074-37)

ELIGIBILITY:
Inclusion Criteria:

* subject whose MDD are single or recurrent without psychotic features according to DSM-IV-TR
* subject with a diagnosis of resistant major depression (≥1 failed antidepressant treatments for the current depressive episode)
* HDRS-21 score ≥ 21
* drug treatment by SSRIs or SNRIs for unipolar patients or with Lithium for bipolar patients for at least 4 weeks
* right-handed patients
* without severe progressive somatic pathology (especially tumor diseases, degenerative diseases)
* without severe cognitive impairment making psychometric evaluation impossible
* excepted antidepressant or Lithium treatment, psychotropic following are tolerated during the course of the study : hydroxyzin; cyamemazin (up to 100 mg/day) ; hypnotics (imidazopyridin).

Exclusion Criteria:

* subject treated with antipsychotics or mood stabilizers or anticonvulsants or by ECT or rTMS for the current depressive episode
* subject resistant to SSRIs or SNRIs for unipolar patients or with Lithium for bipolar patients
* subject with mixed features
* pregnancy and/or lactation
* presence of a specific contraindication for tDCS (e.g., personal history of epilepsy, metallic head implant, cardiac pacemaker)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-07-19 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
change from baseline in HDRS-21 scale | baseline, 1 wk, 2 wk, 4wk, 12 wk, 24 wk
  The changes in HDRS-21 will constitute the major research outcome measure used to assess response to tDCS. Response to treatment is defined as a ≥ 50% reduction in the scores of the HDRS. Remission is defined as a HDRS score ≤ 8.

SECONDARY OUTCOMES:
Change from baseline in MADRS, BDI, HAMA, STAI, YMRS | baseline, 1 wk, 2 wk, 4wk, 12 wk, 24 wk
  Montgomery and Asberg Depression Rating Scale (MADRS) Beck Depression Inventory-13 (BDI) Subscores for anxiety depression scale from HDRS-21 State-Trait Anxiety Inventory (STAI) Young Mania Rating Scale (YMRS) : only for bipolar patient
Change from baseline in COT, TMT, IST and Cardebat fluency task | baseline, 4wk
  Crossing of test (COT) Trail Making test (TMT) Isaacs Set Test (IST) Cardebat fluency task

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel HAFFEN, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (6):
- France (6):
  - CHRU Besancon - Service de Psychiatrie - Centre Investigation Clinique Innovation Technologique (CIC-IT808), Besançon
  - CHU Grenoble - Clinique de Psychiatrie de l'Adulte, Grenoble
  - CH Le Vinatier - Service de Psychiatrie, Lyon
  - Centre Hospitalier Guillaume Régnier - Rennes - Service Hospitalo-Universitaire de Psychiatrie, Rennes
  - Hôpital Civil de Strasbourg - Service de Psychiatrie, Strasbourg
  - Etablissement Public de Santé Mentale - Unité de Recherche Clinique, Ville Evrard

IPD SHARING:
Plan to Share IPD: No